CLINICAL TRIAL: NCT04951973
Title: Comparison of Deep Learning Based Early Warning Score and Conventional Screening System in Rapid Response Team Activation in General Ward Patients
Brief Title: Deep Learning Based Early Warning Score in Rapid Response Team Activation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); VUNO Inc. (Industry); Inha University Hospital (Other); Mediplex Sejong Hospital, Incheon (Unknown); Sejong General Hospital (Other); Dong-A University (Other)
Responsible Party: Sponsor
Other Study IDs: DEWS_2021
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Hospital Rapid Response Team; Hospital Medical Emergency Team
Keywords: deep learning based early warning score; rapid response team; in-hospital cardiac arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Deep Learning Based Early Warning Score (DEWS) — DEWS use 4 vital signs (systolic blood pressure, HR, respiratory rate, and body temperature) to predict in-hospital cardiac arrest. Deep-learning approach facilitates learning the relationship between the vital signs and cardiac arrest to achieve the high sensitivity and low false-alarm rate of the track-and-trigger system (TTS).

SUMMARY:
The objective of this study is to evaluate the safety and clinical usefulness of the Deep learning based Early Warning Score (DEWS).

DETAILED DESCRIPTION:
SPTTS is the representative trigger tracking system. In addition to the conventional SPTTS, DEWS will be calculated at each time point by the previously developed algorithm. SPTTS and DEWS will be shown simulataneously on the screening board. The rapid response team performs the rescue activity as before, using both SPTTS and DEWS simultaneously.

The alarm threshold setting of DEWS will be changed to 70 points, 75 points, and 80 points every month.

The primary and secondary outcomes will be evaluated to compare SPTTS and DEWS (based on each threshold).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to general ward and monitored by in-hospital rapid response system

Exclusion Criteria:

* patients admitted to pediatric ward
* patients in emergency room, intensive care unit, and operating room

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to general ward
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
In-hospital cardiac arrest | 3 month
  Compare the predictability of in-hospital cardiac arrest between DEWS and SPTTS.

SECONDARY OUTCOMES:
Alarm coincidence | 3 month
  Evaluate the alarm coincidence between DEWS and SPTTS.
Total alarm count. | 3 month
  Compare the total alarm count between DEWS and SPTTS.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon JM, Lee Y, Lee Y, Lee S, Park J. An Algorithm Based on Deep Learning for Predicting In-Hospital Cardiac Arrest. J Am Heart Assoc. 2018 Jun 26;7(13):e008678. doi: 10.1161/JAHA.118.008678. PMID 29945914
- [Background] Cho KJ, Kwon O, Kwon JM, Lee Y, Park H, Jeon KH, Kim KH, Park J, Oh BH. Detecting Patient Deterioration Using Artificial Intelligence in a Rapid Response System. Crit Care Med. 2020 Apr;48(4):e285-e289. doi: 10.1097/CCM.0000000000004236. PMID 32205618
- [Derived] Cho KJ, Kim JS, Lee DH, Lee SM, Song MJ, Lim SY, Cho YJ, Jo YH, Shin Y, Lee YJ. Prospective, multicenter validation of the deep learning-based cardiac arrest risk management system for predicting in-hospital cardiac arrest or unplanned intensive care unit transfer in patients admitted to general wards. Crit Care. 2023 Sep 5;27(1):346. doi: 10.1186/s13054-023-04609-0. PMID 37670324